CLINICAL TRIAL: NCT01753453
Title: A Pilot, Exploratory, Randomized, Phase 2 Safety Study Evaluating Tumor Cell (Plasma Cell) Mobilization and Apheresis Product Contamination in Plerixafor Plus Non-pegylated G-CSF Mobilized Patients and in Non-pegylated G-CSF Alone Mobilized Patients
Brief Title: An Exploratory Safety Study to Investigate the Extent of Tumor Cell Mobilization (TCM) After Use of G-CSF Alone or G-CSF Plus Plerixafor in Multiple Myeloma (MM) Patients Who May be Poor Mobilizers of Stem Cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARD12858; MOZ23510 (Other: Genzyme); 2011-004783-30 (EudraCT Number)
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Multiple Myeloma
Keywords: Hematopoietic stem cell transplantation; Tumour cell mobilization
MeSH Terms: conditions — Multiple Myeloma | interventions — plerixafor; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-CSF alone (Active Comparator): Patients will receive G-CSF for 5 consecutive days
  Interventions: Drug: Granulocyte-colony stimulating factor (G-CSF)
- G-CSF plus plerixafor (Experimental): Patients will receive G-CSF for 4 consecutive days, then receive plerixafor before the 5th dose of G-CSF
  Interventions: Drug: Plerixafor; Drug: Granulocyte-colony stimulating factor (G-CSF)

INTERVENTIONS:
Drug: Plerixafor — 240mcg/kg, solution, subcutaneous injection
  Other Names: Mozobil,AMD3100
  Arms: G-CSF plus plerixafor
Drug: Granulocyte-colony stimulating factor (G-CSF) — 10 mcg/kg, solution, subcutaneous injection

SUMMARY:
The primary objective of this study is to evaluate tumor cell mobilization (TCM) with non-pegylated G-CSF alone compared with non-pegylated G-CSF plus plerixafor in patients with multiple myeloma (MM) who are potentially poor mobilizers of hematopoietic stem cells (HSC).

Second objectives are to evaluate survival and disease status of G-CSF alone compared with GCSF plus plerixafor, and the efficacy and safety of G-CSF plus plerixafor when used to mobilize stem cells for autologous transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of MM in partial response or complete response, who are undergo an autologous hematopoietic stem cell transplantation and could be considered potentially poor mobilizers.

Exclusion Criteria:

* Does not have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Has a history of any acute or chronic leukemia (including myelodysplastic syndrome).
* Had prior allogeneic or autologous transplantation.
* Less than 3 to 6 weeks since last anti-cancer therapy.
* Chemotherapy for mobilization is not allowed.
* Has bone marrow involvement >10% assessed based on the most recent bone marrow aspirate or biopsy performed prior to first dose of G-CSF.
* Was treated with G-CSF or other cytokine within 14 days prior to the first dose of G-CSF for mobilization.
* Has previously received plerixafor.
* Is known to be HIV positive.
* Has active hepatitis B or hepatitis C.
* Has an acute infection within 24 hours prior to dosing or antibiotic therapy within 7 days prior to the first dose of G-CSF.
* Has hypercalcaemia as evidenced by >1 mg/dL above upper limit of normal (ULN).
* Previously received investigational therapy within 4 weeks of screening in this protocol or currently enrolled in another investigational protocol during the mobilization phase.
* Has central nervous system involvement including brain metastases or leptomeningeal disease.
* Has an electrocardiogram (ECG) or study result indicative of cardiac ischemia or a history of clinically significant rhythm disturbance(arrhythmias), or other conduction abnormality.
* Has co-morbid condition(s), which may render the patient at high risk from treatment complications or impairs his/her ability to comply with the study treatment and protocol.
* Has a white blood cell (WBC) count <2.5 x 10^9/L.
* Has an absolute neutrophil count (ANC) <1.5 x 10^9/L.
* Has a platelet count <100 x 10^9/L.
* Has an estimated creatine clearance ≤50 mL/min.
* Has aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT), alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT), and total bilirubin ≥2.5 x ULN.
* Does not have adequate cardiac, and pulmonary function sufficient to undergo apheresis and transplantation.
* Pregnant or breastfeeding women.
* Does not agree to use a highly effective method of contraception while on study treatment and for at least 3 months following study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The presence of myeloma tumor cells as measured by the percentage of myeloma tumor cells/CD34+ cells | Day 1 to Day 8 of the apheresis/treatment period
  Peripheral blood parameters
The presence of myeloma tumor cells as measured by the percentage of myeloma tumor cells/plerixafor cumulative dose/kg body weights | Day 5 to Day 8 of the apheresis/treatment period
  Peripheral blood parameters
The presence of myeloma tumor cells as measured by the percentage of myeloma tumor cells/G-CSF cumulative dose/kg body weight | Day 5 to Day 8 of the apheresis/treatment period
  Peripheral blood parameters
The change in tumor cell mobilization(TCM) in the peripheral blood | Day 4 pre-G-CSF to Day 5 pre-G-CSF
  Peripheral blood parameters
The number of myeloma tumor cells per patient at each apheresis | Day 1 to Day 8 of the apheresis/treatment period
  Apheresis product parameters
The number of patients who mobilize at least 4.5x10^5 myeloma tumor cells/kg body weight as measured in each apheresis product | Day 5 to Day 8 of the apheresis/treatment period
  Apheresis product parameters

SECONDARY OUTCOMES:
CD34+ stem cell yield in the apheresis product | Day 1 to Day 8 of the apheresis/treatment period
The number of patients that proceed to transplantation | Up to 2 months after final apheresis
Overall survival | Day 100 post transplant and up to 2 years post first-G-CSF dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- Investigational Site Number 056002, Bruges, Belgium
- Investigational Site Number 233001, Tallinn, Estonia
- Investigational Site Number 440001, Vilnius, Lithuania
- Sweden (2):
  - Investigational Site Number 752001, Stockholm
  - Investigational Site Number 752002, Umeå